CLINICAL TRIAL: NCT01287819
Title: Polymorphisms of Apolipoprotein E Gene and the Presentation of Resting-state Functional MRI
Brief Title: Apolipoprotein E Gene and Functional MRI
Acronym: fMRI
Status: Completed | Type: Observational
Sponsor: Taipei Medical University Shuang Ho Hospital (Other)
Collaborators: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Chaur-jong Hu, Chief of Neurology department, Taipei Medical University Shuang Ho Hospital
Other Study IDs: CRC-12-10-04
Record Dates: First submitted 2011-01-31; First posted 2011-02-01 (Estimated); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — DNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- APOE4 (+) and APE4 (-): APOE4 (+) 10 people APOE4 (-) 20 people from 200 participants

SUMMARY:
1. Apolipoprotein E gene (ApoE) is the most important genetic factor for Alzheimer disease (AD) and an important genetic factor for outcome of brain injury situations.
2. Function magnetic resonance imaging (fMRI) is a powerful tool for study of both brain regional functions and brain network.
3. Study about genetic contribution on fMRI is an emerging concept, which will help on understanding about how the genetics affecting the brain function.

DETAILED DESCRIPTION:
There are about 4-10% people aged and over 65 years suffering from dementia in Taiwan. Dementia caused by diverse diseases, including Alzheimer's disease (AD), fronto-temporal dementia (FTD), dementia with Lewy body (DLB), Parkinson's disease dementia (PDD) and vascular dementia (VaD), is a neurodegenerative disease characterized by memory impairment, cognitive dysfunctions, behavioral disturbances and various kinds of psychiatric manifestations. AD is the most common cause of dementia in the world. Although the real pathophysiology of AD is still obscure, the compelling evidence has shown genetic factor should play an important role in the occurrence of AD. There are three genes, in terms of amyloid precursor protein (APP), presenilin-1 (PS1) and presenilin-2 (PS2), linked in the familial AD. Mutations on these genes would result in familial AD, which account for only less than 5% of AD. The only one well-documented genetic risk factor for sporadic AD is apolipoprotein E, ε4 allele (ApoE4). ApoE gene contains three genetic polymorphisms, ε2, 3, 4 and ApoE4 has been found associated with many brain injury situations, such as poor outcome for traumatic brain injury (TBI), Parkinson disease dementia (PDD). These findings might support ApoE to be important for brain functions but the real mechanisms remain further clarification. Functional magnetic resonance imaging (fMRI) is a powerful tool for study of both brain regional functions and brain network. To our knowledge, only few reports in top journals indicated genetic background is an important contributor for fMRI presentations. This could be a new filed of neuroscience. In this study, we will explore whether ApoE genetic polymorphisms affect the presentation of fMRI and realize some functions of ApoE in the brain. In addition, our data could enhance the new concept about the association between genetics and brain function.

ELIGIBILITY:
Inclusion Criteria:

* people aged 45-65 years without cognitive impairment

Exclusion Criteria:

* unable to take APOE genotyping or undergo functional MRI

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: people aged 45-65 years taking health examination in TMU SHH no cognitive impairment by MMSE and AD8 screening
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2012-05; Primary Completion 2013-04-17 (Actual); Study Completion 2013-04-18 (Actual)

PRIMARY OUTCOMES:
amyloid load by amyloid-PET examination | every 5 years
  The primary end point of this study is the quantity of amyloid load in brain. The amyloid load will be calculated based on the results of AV45 PET study. The comparison between mTBI and controls will be conducted by ANOVA test. The confounders include vascular risks for AD, such as hypertension, diabetes, and APOE genotypes, education.

CONTACTS AND LOCATIONS:
Overall Officials: Chaur-Jong Hu, M.D., Principal Investigator — Taipei Medical University Shuang Ho Hospital
Locations (1):
- Chaur-Jong Hu, New Taipei City, Taiwan

REFERENCES:
- [Derived] Chen CJ, Chen CC, Wu D, Chi NF, Chen PC, Liao YP, Chiu HW, Hu CJ. Effects of the apolipoprotein E epsilon4 allele on functional MRI during n-back working memory tasks in healthy middle-aged adults. AJNR Am J Neuroradiol. 2013 Jun-Jul;34(6):1197-202. doi: 10.3174/ajnr.A3369. Epub 2012 Dec 28. PMID 23275593